CLINICAL TRIAL: NCT04194697
Title: A Study to Assess Effect of Exercise Program Provided by Smartphone Application on the Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4646-CL-0001
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Exercise program; Smartphone application
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants will conduct exercise programs provided by the app 3 times a week for 12 weeks. Except for the exercise program provided by the app, the amount of activity and exercise in daily life will not change from before the study.
  Interventions: Behavioral: Exercise
- Non-exercise group (Other): Participants will not change the amount of activity or exercise in daily life from before the study.
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise program
  Arms: Exercise group
Behavioral: No exercise — No exercise program
  Arms: Non-exercise group

SUMMARY:
The primary objective of this study is to explore the effect of an exercise program combining aerobic and resistance exercises provided by mobile healthcare applications (hereinafter referred to as "app") on the body composition in app-using exercise group compared to non-exercise group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can perform a 12-week exercise program using the specified app during the study in Japan if they are assigned to the app-using exercise group.
* Subjects who agree to perform a 12-week exercise program using the app during the period specified in the protocol and not to change activities/exercise of daily living compared with before participation in the study except for the exercise program using the app if they are assigned to the app-using exercise group, or subjects who agree not to change activities/exercise of daily living compared with before participation in the study during the period specified in the protocol if they are assigned to the non-exercise group.
* Subjects with body mass index (BMI) of 25.0 kg/m^2 or more and less than 30.0 kg/m^2 at screening and baseline
* Subjects with waist circumferences meeting the following at screening and baseline. Male: 85 cm or more, Female: 90 cm or more
* Female subject who applied to one of the following

  * Subjects who are postmenopausal (without a menstrual period for at least 1 year) at the time of informed consent.
  * Subjects of non-childbearing potential due to undergoing surgery.
  * Females of childbearing potential who agree to use contraception during the participation in the study and have a negative pregnancy test at screening and baseline.
* Subjects who agree not to participate in clinical studies of drugs, regenerative medicine products, or medical devices, post-marketing clinical studies, or clinical research (including studies that do not use drugs, regenerative medicine products, or medical devices as with this study) other than this study after providing informed consent until the completion of the examination/observation at Week 12.

Exclusion Criteria:

* Subjects who regularly perform at least 1 session of exercise per week for at least 30 minutes per session on average other than activities of daily living during 6 months before providing informed consent.
* Subjects who receive treatment for obesity on an outpatient basis at the time of informed consent or plan to start treatment for obesity on an outpatient basis during the period until the completion of the examination/observation at Week 12.
* Subjects whose systolic blood pressure (sitting position at rest) is 160 mmHg or more or whose diastolic blood pressure (sitting position at rest) is 100 mmHg or more at screening or baseline.
* Subjects with concomitant uncontrolled hypertension or concomitant hypertension that is considered likely to be exacerbated by the exercise intervention.
* Subjects with previous or concomitant severe heart diseases (ischemic heart disease, myocardial infarction, congestive heart failure, angina pectoris, and arrhythmia requiring treatment with β-blockers and other drugs, etc.).
* Subjects with previous or concomitant cerebrovascular disorders (cerebral infarction, transient cerebral ischemia, etc.).
* Subjects with fasting blood glucose of 250 mg/dL or more or with positive urinary ketone bodies at screening.
* Subjects with concomitant uncontrolled diabetes or with diabetic complications (diabetic neuropathy, diabetic nephropathy, and diabetic retinopathy excluding simple retinopathy).
* Subjects with concomitant retinal neovascular lesions (exudative age-related macular degeneration, retinal vein occlusion, etc.) or concomitant retinopathy occurring within 6 months after laser photocoagulation.
* Subjects with previous or concomitant arteriosclerosis obliterans of lower extremities
* Subjects with concomitant motor disorders.
* Subjects with concomitant severe respiratory diseases.
* Subjects with concomitant severe liver diseases (viral hepatitis, drug-induced liver injury, etc.).
* Subjects with concomitant severe renal diseases (acute renal failure, glomerulonephritis, interstitial nephritis, etc.).
* Subjects with previous or concomitant malignancies. However, subjects are allowed to be enrolled if they have experienced no recurrence without the need for treatment within 5 years before providing informed consent.
* Subjects with previous or concomitant schizophrenia, psychiatric disorders such as bipolar disorder or major depressive disorder, or dementia.
* Subjects who are taking any of the following drugs at the time of informed consent: insulin preparations, sulfonyl urea hypoglycemic agents, short-acting insulin secretagogues (glinide), Glucagon-like peptide (GLP)-1 receptor agonists, biguanides, thiazolidines, Sodium-glucose co-transporter (SGLT)2 inhibitors, and anti-obesity drugs, or subjects who plan to receive any of these drugs during the period until the completion of the examination/observation at Week 12.
* Subjects who are taking any of the following at the time of informed consent: antidyslipidemic agents or drugs affecting lipid metabolism, supplements, and health foods (including foods for specified health use and foods with functional claims), or subjects who plan to take any of these during the period until the completion of the examination/observation at Week 12. However, subjects are allowed to take these drugs, supplements, or foods if they can take them with a stable dosage from at least 28 days before baseline until the completion of the examination/observation at Week 12.
* Subjects who have metal placed by lumbar spinal surgery and other surgery at the site where abdominal CT scan is performed.
* Subjects with implantable medical devices such as cardiac pacemakers and implantable defibrillators.
* Subjects who have participated or are participating in clinical studies of other drugs, regenerative medicine products, or medical devices, post-marketing clinical studies, or clinical research (including studies that do not use drugs, regenerative medicine products, or medical devices as with this study) within 12 weeks (84 days) before screening.
* Subjects who are employed by the research implementing entity of this study or institutions/organizations related to this study.
* Subjects who are considered ineligible for the participation in this study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visceral fat area | Baseline and Week 12
  Visceral fat area will be measured with computed tomography (CT).
Change from baseline in body fat ratio | Baseline and Week 12
  Total fat ratio will be derived from body composition analyzer.

SECONDARY OUTCOMES:
Change from baseline in subcutaneous fat area | Baseline and Week 12
  Subcutaneous fat area will be measured with CT.
Change from baseline in total fat area | Baseline and Week 12
  Body fat area will be measured with CT.
Change from baseline in muscle mass | Baseline and Week 12
  Muscle area will be measured with body composition analyzer.
Change from baseline in waist circumference | Baseline and Week 12
  Waist circumference will be measured with measuring tape.
Change from baseline in body weight | Baseline and Week 12
  Body weight will be measured with body composition analyzer.
Number of participants with Adverse Events (AEs) | Up to Week 12
  An adverse event is any untoward medical occurrence in subjects, which does not necessarily have to have a causal relationship with this study.
  An event that meets either "possibly related" or "probably related" is defined as "an adverse event whose causal relationship with this study cannot be ruled out" or "an adverse event whose causal relationship with the exercise intervention cannot be ruled out."

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Inc., Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Toshima-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.